CLINICAL TRIAL: NCT06767605
Title: Registro Español de Enfermedades Hepáticas Colestásicas y Autoinmunes (ColHai)
Brief Title: Spanish Registry of Autoimmune and Cholestatic Liver Diseases (ColHai)
Acronym: ColHai
Status: Recruiting | Type: Observational
Sponsor: Asociación Española para el Estudio del Hígado (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2016/0565
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis Autoimmune Disease; Primary Biliary Cholangitis (PBC); Primary Sclerosing Cholangitis (PSC); Cholestatic Genetic Diseases
Keywords: Cholestatic Genetic Diseases; Primary Sclerosing Cholangitis (PSC); Hepatitis Autoimmune Disease; Primary Biliary Cholangitis (PBC); PFIC tipo 1; PFIC tipo 2; PFIC tipo 3; PFIC tipo 4; BRIC tipo 1; BRIC tipo 2; Alagille syndrome; Rotor syndrome; Dubin Johnson syndrome; Genetic disease; Registry; cholestatic diseases
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Cholangitis, Sclerosing; Alagille Syndrome; Hyperbilirubinemia, Hereditary; Jaundice, Chronic Idiopathic; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 35 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the registry is to know the status of primary biliary colgantis, autoimmune hepatitis, primary sclerosing cholagitis and genetic cholestatic diseases in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis for PBC, HAI, PSC, genetic cholestatic disease

Exclusion Criteria:

* Refusal to sign the informed consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis for PBC, HAI, PSC or any genetic cholestasis
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence and characteristics of autoimmune and cholestatic liver disease in Spain | 2025
  Evaluation of clinical characteristics of autoimmune and cholestatic liver diseases

SECONDARY OUTCOMES:
Development of liver-related events in autoimmune ahd cholestatic liver diseases | 2025
Treatment of autoimmune and cholestatic liver diseases in Spain | 2016-2030

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carlota Londoño Londoño, Study Director — Asociación Española para el Estudio del Hígado
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No